CLINICAL TRIAL: NCT02849548
Title: Can Blocking the Orexin System Enhance Sleep's Benefits to Therapeutic Exposure for PTSD?
Brief Title: Suvorexant and Sleep's Benefits to Therapeutic Exposure for Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Howard University (Other)
Collaborators: Georgetown-Howard Universities Center for Clinical and Translational Science (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GHUCCTS2016-0377; 1K01MH110647-01A1 (NIH)
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- suvorexant (Experimental): 10 to 20 mg to be administered after an evening written trauma narrative exposure session.
  Interventions: Drug: suvorexant
- Placebo pill (Placebo Comparator): A pill without active ingredients
  Interventions: Other: placebo

INTERVENTIONS:
Drug: suvorexant — First in class orexin antagonist approved by the FDA for the treatment of insomnia
  Other Names: Belsomra
  Arms: suvorexant
Other: placebo — Pill with inactive ingredients
  Arms: Placebo pill

SUMMARY:
The purpose of this study is to examine effects of blocking the orexin system with suvorexant after exposure-based intervention for posttraumatic stress disorder (PTSD) on sleep, PTSD symptoms, and intersession habituation.

DETAILED DESCRIPTION:
Cognitive behavioral therapies (CBT) that include exposure to trauma memories are considered first line treatments for PTSD. However, approximately 1/3 of patients who complete CBT for PTSD do not achieve remission, and hyperarousal symptoms including sleep disturbances are less responsive to CBT than other PTSD symptoms. Despite these limitations, CBT outcomes are generally superior to outcomes of pharmacotherapy. It is, therefore, imperative to identify strategies to improve effectiveness of treatments for PTSD, particularly hyperarousal symptoms.

Disturbed sleep is common in PTSD. Studies of PTSD and anxiety and mood disorders have shown that impaired sleep before psychotherapy predicted less favorable responses. Sleep has been implicated in learning processes that are a key to adaptive processing of trauma memories such as extinction learning and generalization of extinction. Our recent PTSD study showed that preserved slow-wave sleep (SWS), less increase in rapid-eye-movement (REM) density, and reduced wake after sleep onset (WASO) during sleep following an evening session of written narrative exposure (WNE: writing about one's traumatic experience) was associated with greater PTSD symptom reduction. These findings suggest that increased nocturnal arousal compromises sleep's benefits to emotional processing of trauma memories. Identifying strategies to reduce nocturnal arousal and promote sleep characteristics associated with emotional adaptation could enhance PTSD treatment outcomes.

Orexins are neuropeptides implicated in regulating both sleep/wakefulness and emotional behaviors, including anxiety. Inhibiting the orexin system promoted slow-wave patterns and reduced wake in animal models. The first orexin receptor antagonist (suvorexant) was recently approved for treatment of insomnia. Suvorexant reduced WASO and latency to persistent sleep and increased SWS and REM sleep in humans with insomnia. In addition, administrations of orexin-A increased anxiety-like behaviors in rodents, and administrations of an orexin receptor-1 antagonist to mice facilitated extinction of conditioned fear, an animal model of recovery from PTSD and anxiety disorders.

Objective: To examine effects of blocking the orexin system with suvorexant after WNE on sleep, PTSD symptoms, and intersession habituation.

The investigators will utilize the WNE paradigm in which participants with PTSD write about their traumatic experiences in the evening and morning sessions with intervening sleep. Suvorexant or placebo will be administered after the evening WNE, and sleep will be recorded.

The investigators hypothesize that 1) Suvorexant will promote the sleep characteristics that have been associated with more favorable treatment outcomes and emotional adaptation (e.g., increased SWS and REM sleep, reduced WASO) compared with placebo; 2) Participants given suvorexant will have greater PTSD symptom reduction and intersession habituation indexed by reduction of maximum pulse rate compared with participants given placebo; and 3) The greater PTSD symptom reduction and intersession habituation in the suvorexant group will be accounted for by effects of the medication on sleep.

ELIGIBILITY:
Inclusion Criteria:

- Adult men and women (age 18 or older) who meet the Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for PTSD.

Exclusion Criteria:

* Medical or psychiatric conditions that require consistent use of medication that affects sleep or psychiatric symptoms, except for hormonal contraceptives
* Any persistent medical condition that affects sleep
* Inability to remember most details of the index event
* Diagnosis of a sleep disorder other than insomnia including polysomnography findings of apnea/hypopnea index > 10/hour
* Consumption of more caffeine than 5 cups of coffee/day equivalent
* Smoking > 20 cigarettes/day
* Habitual bedtimes after 3AM, habitual rise times after 10AM, or average napping > 2 hour/day in a given week
* Moderate or severe alcohol use disorder within the past 6 months or moderate or severe drug use disorder within the past year
* Positive urine toxicology for illicit drugs including cannabis
* A history of psychotic disorders or bipolar disorder
* Current depression with history of recurrent depression that precedes exposure to a traumatic event
* Suicidal ideation with intent to act or with specific plan and intent in the past 6 months [Type 4 - 5 ideation on the Columbia Suicide Severity Rating Scale (C-SSRS)] or history of a suicide attempt
* Completion of exposure-based therapy targeting the index trauma
* Pregnancy or breast feeding
* Known sensitivity or allergy to an orexin receptor antagonist
* Limited ability to read or write English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ihori Kobayashi, Ph.D., Principal Investigator — Howard University
Locations (1):
- Clinical Research Unit; Howard University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified final dataset will include scores/values obtained through self-report survey, interviews, narrative writing, pulse recording, and polysomnography. Even though personally identifiable information will be removed from the final dataset, there remains the possibility that participants' identities are deduced from information about their traumatic events. Therefore, participants' trauma narratives and details of traumatic events disclosed during the writing sessions and interviews will not be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available after the first publication is published.
Access Criteria: Given the highly sensitive nature of the data which includes participants' mental and physical health information, we will make the de-identified data available to users only under a data-sharing agreement that: 1) the data will be used only for research purposes; 2) users will not identify any individual participant; 3) users utilize appropriate computer technology to ensure data security; and 4) users destroy or return the data after analyses are completed.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suvorexant | Placebo Pill
Started | 13 | 14
Completed | 11 | 12
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant | Placebo Pill | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (8) | 35 (10) | 33.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 11 | 13 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 5 | 7 | 12
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27
1-week Clinician Administered PTSD Scale for DSM-5 (CAPS-5) [Mean (Standard Deviation); unit: units on a scale] — A structured clinical interview used to assess posttraumatic stress disorder (PTSD) symptom severity for the preceding week. Items are scored on a 5-point scale, and a total score is obtained by summing the 20 symptom items, with higher scores indicating greater PTSD symptom severity. The total scores range from 0 - 80.
  units on a scale | 23.2 (7.8) | 28.0 (12.4) | 25.7 (10.5)
Baseline-corrected highest SUDS at the 1st written narrative exposure session [Mean (Standard Deviation); unit: units on a scale] — The subjective unit of distress scale (SUDS) is a numerical scale that is administered orally. It ranges from 0 - 100 in which 0 indicates no stress at all, and 100 indicates the highest stress level. The highest SUDS score for each session was identified and corrected for the baseline SUDS of the session by subtracting the baseline SUDS from the SUDS within the session; therefore, the baseline-corrected SUDS scores can range from 0 to 100.
  units on a scale | 32.0 (18.4) | 35.3 (18.3) | 33.7 (18.1)
Baseline-corrected highest 2-min average pulse rate at the 1st written narrative exposure session [Mean (Standard Deviation); unit: beats per minute] — The average pulse rate for a 5-minute baseline and each 2-minute epoch during 30-min written narrative exposure were computed. The highest average pulse rate for each session was identified and corrected for the baseline pulse rate of the session by subtracting the baseline average pulse rate from the highest average pulse rate within the session. The Baseline-corrected highest pulse rate values reported here are small because the baseline average pulse rate of the session was subtracted from the highest 2-minute average pulse rate of the session.
  beats per minute | 5.9 (4.6) | 7.2 (5.9) | 6.6 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: The Clinician Administered PTSD Scale for DSM-5 (CAPS-5) Score at Week 2
Description: A structured clinical interview used to assess posttraumatic stress disorder (PTSD) symptom severity for the preceding week. Items are scored on a 5-point scale, and a total score is obtained by summing the 20 symptom items, with higher scores indicating greater PTSD symptom severity. The total scores range from 0 - 80.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo Pill
Number analyzed (Participants) | 11 | 12
score on a scale | 16.6 (7.3) | 17.1 (12)

2. Secondary Outcome: The Baseline-corrected Highest Subjective Unit of Distress Scale (SUDS) Scores at the Last Written Narrative Exposure Session
Description: The subjective unit of distress scale (SUDS) is a numerical scale that is administered orally. It ranges from 0 - 100 in which 0 indicates no stress at all, and 100 indicates the highest stress level. The highest SUDS score for each session was identified and corrected for the baseline SUDS of the session by subtracting the baseline SUDS from the SUDS within the session; therefore, the baseline-corrected SUDS scores can range from 0 to 100.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo Pill
Number analyzed (Participants) | 11 | 12
score on a scale | 18.9 (15.8) | 40.3 (22.0)

3. Secondary Outcome: The Baseline-corrected Highest Pulse Rate Across at the Last Written Narrative Exposure Session
Description: The average pulse rate for a 5-minute baseline and each 2-minute epoch during 30-min written narrative exposure were computed. The highest average pulse rate for each session was identified and corrected for the baseline pulse rate of the session by subtracting the baseline average pulse rate from the highest average pulse rate within the session. The Baseline-corrected highest pulse rate values reported here are small because the baseline average pulse rate of the session was subtracted from the highest 2-minute average pulse rate of the session.
Time Frame: 1week
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Suvorexant | Placebo Pill
Number analyzed (Participants) | 11 | 12
beats per minute | 5.3 (3.0) | 4.8 (2.4)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Interview with open-ended questions.
Arm/Group | Suvorexant | Placebo Pill
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 9/13 | 9/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Suvorexant (N=13) | Placebo Pill (N=14)
Fatigue (General disorders) | 4 | 3
Somnolence (Nervous system disorders) | 3 | 2
Depression (Nervous system disorders) | 2 | 1
Anxiety (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 2
Nightmare (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT02849548/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT02849548/SAP_001.pdf